CLINICAL TRIAL: NCT02782299
Title: Shared Decision Making in Older Adults With Distal Radius Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB closed project as the continuing review was not submitted. PI has left WU.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201512001
Record Dates: First submitted 2016-05-01; First posted 2016-05-25 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Radius Fracture
Keywords: Decision aid; Shared decision making; Older adult patients; Distal radius fracture
MeSH Terms: conditions — Radius Fractures; Wrist Fractures | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): This group will not be exposed to the decision aid. Patients will complete the same surveys, and will be followed for the same length of time.
- Decision Aid (Experimental): This group will be exposed to the decision aid before the patients appointment with the surgeon. Patients will also complete the same outcome surveys, and will be followed for the same length of time.
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Decision Aid — Decision aid which is still under revision will include unbiased information to assist is clarifying values and informing patients with distal radius fractures.
  Arms: Decision Aid

SUMMARY:
This is a study to investigate the use of a Decision Aid for shared decision making in older adults with distal radius fractures. The goal is to improve patient decisions making, and improve patient knowledge through the use of a validated decision aid.

DETAILED DESCRIPTION:
Shared decision making has become a increasingly important with the goal of helping patients make decisions that more align with patients values and goals. Decision aids are validated instruments that provide unbiased information and guide patients through questions that allow patients to clarify patients goals.

Older adults with distal radius fractures have increasing evidence of ability to tolerate residual deformity with little to no functional deficits, which has called into question the indications for surgery. In situations where the operative indications are not clear, it is important to engage the patient in the risk and benefits of the decision.

This trial is a prospective trial with two groups, one standard of care, and one with the decision aid.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture within the past 2 weeks
* Initial appointment seeing Attending
* Age 65+

Exclusion Criteria:

* Non english speaker
* Dementia or other mental limitation preventing ability to complete survey
* Other traumatic injuries in extremity that would affect surgical decision

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Decision Conflict Score | Immediate post appointment
  Validated measure for decision conflict

SECONDARY OUTCOMES:
Decision regret scale | 6 weeks and 6 months post appointment
  Validated measure for decision regret
Patient knowledge | immediate post appointment
  Knowledge quiz created to evaluate knowledge of distal radius treatment options

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Calfee, MD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University-St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No